CLINICAL TRIAL: NCT06590922
Title: Application of New Oropharyngeal Airway Management in Obese Patients Undergoing Painless Gastroenteroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Wu, chief physician, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YXLL-KY-2024 (082)
Record Dates: First submitted 2024-09-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Gastrointestinal Endoscopy; Airway Management
MeSH Terms: conditions — Obesity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using a new oropharyngeal airway set (Experimental): Prior to induction of anesthesia and until the end of the gastroenteroscopy, oxygen was continuously supplied through a catheter partially attached to the endoscopic bite.
  Interventions: Device: Group using new oropharyngeal airway (experimental group)
- The conventional endoscopic bite group (Active Comparator): Oxygen was administered continuously through a common nasal catheter until the end of the gastroenteroscopy prior to induction of anesthesia
  Interventions: Device: The conventional endoscopic biting group (control group)

INTERVENTIONS:
Device: Group using new oropharyngeal airway (experimental group) — Before anesthesia induction, study participants in the experimental group received 5-6L/min oxygen for about 1min through an endoscopic bite oxygen supply device, and anesthesia induction was administered with propofol 3mg/kg and sufentanil 7μg.Sufentanil was given at the beginning of pre-oxygen inhalation, and propofol was given 1min later. When participants achieved sufficient sedation (about BIS40), they were placed into the oropharyngeal airway through the endoscopic bite and began gastroscopy.Anesthetic maintenance was administered with a continuous pump of 5mg/kg·h propofol until completion of the examination.
  Arms: Using a new oropharyngeal airway set
Device: The conventional endoscopic biting group (control group) — Prior to induction of anesthesia, control study participants inhaled 5 to 6L/min of oxygen through a nasal catheter for approximately 1 minute.Anesthesia was induced by propofol 3mg/kg and sufentanil 7μg.Sufentanil was given at the beginning of pre-oxygen inhalation, and propofol was given 1min later. The endoscopic procedure began when the study participants reached sufficient sedation (about BIS40) and the ordinary endoscopic bite group reached sufficient sedation.Anesthetic maintenance was administered with a continuous pump of 5mg/kg·h propofol until completion of the examination.
  Arms: The conventional endoscopic bite group

SUMMARY:
Painless endoscopy is a popular method of endoscopic diagnosis and treatment. Propofol combined with fentanyl general intravenous anesthesia has been widely used in painless endoscopic diagnosis and treatment.However, the combined application of the two has a significant respiratory center inhibition effect, resulting in a decrease in blood oxygen saturation of patients, especially obese patients, who are more likely to suffer from a sudden drop in blood oxygen and even threaten their lives .Due to the potential risk of upper airway obstruction in some obese patients, intraoperative hypopnea may occur during painless colonoscopy due to the influence of sedative and analgesic drugs, resulting in hypoxia in patients. In addition, the anatomical and pathological changes of obese patients themselves make hypoxia tolerance poor and airway establishment difficult, which may endanger the safety of patients .Currently, there is no special oropharyngeal ventilation device used during gastroenteroscopy. Recently, a new type of oropharyngeal ventilation channel has been developed and applied in clinic.Compared with the conventional nasal catheter, the new oropharyngeal airway nasal mask can better fit the patient's face, ensure the air tightness inside the nose mask and maximize the oxygen supply efficiency. The carbon dioxide outlet connected to the oropharyngeal airway body can not only collect the patient's exhaled gas, but also reduce the backflow of carbon dioxide gas.It can also access carbon dioxide detection equipment to monitor the patient's PCO2 at the end of breath in real time .In order to evaluate whether the new oropharyngeal airway can reduce the incidence of hypoxia in ordinary patients during painless gastroenteroscopy, the investigators prepared this study and explored the safety and effectiveness of the new oropharyngeal airway .

DETAILED DESCRIPTION:
1. The study population was recruited by the investigator participating in the clinical trial under the control of the principal investigator. 226 obese patients (30≤BMI≤40) who had undergone painless gastroenteroscopy since the same day were selected and informed and consented to the clinical trial.2. Sample size calculation:According to the pre-test results of obese people, the incidence of hypoxia in the test group and the control group was 0.08 and 0.26, respectively. The sample size was calculated using PASS software, and the bilateral test level α=0.05 was set, and the test efficacy power=0.9 was set. According to the incidence of hypoxia, 90 cases were required in each group, and 113 cases in each group were calculated after considering 20% shedding rate.A total of 226 cases.3. Specific study contents: Study participants entered the examination room to establish venous access, and used 2% lidocaine gel 5ml containing mouthwash and pharynx.Heart rate (HR), pulse oxygen saturation (SpO2), end-expiratory carbon dioxide, ECG monitoring, and non-invasive blood pressure (measured every 2.5 minutes) were routinely monitored before anesthesia induction.Ask patient to lie on left side.In this study, the investigators participating in this clinical trial plan to implement simple randomization using SAS: (1) The group using the new oropharyngeal airway (trial group) : Oxygen is continuously supplied through a catheter partially attached to the endoscopic bite before induction of anesthesia until the end of gastroenteroscopy.(2) In the conventional endoscopic bite group (control group), oxygen was continuously supplied through a common nasal catheter before induction of anesthesia until the end of gastroenteroscopy.The entire trial operation process was completed by the investigators participating in the clinical study.Before induction of anesthesia, study participants in the experimental group received 5-6L/min of oxygen for about 1 minute through an endoscopic biting oxygen supply device, and participants in the control group inhaled 5-6L/min of oxygen for about 1 minute through a nasal catheter.Propofol 3mg/kg and sufentanil 7μg were used to induce anesthesia in both groups.Sufentanil was given at the beginning of pre-oxygen inhalation, and propofol was given 1 minute later. When participants achieved sufficient sedation (BIS40 left and 12 right), the new oropharyngeal airway group was placed into the oropharyngeal airway through the endoscopic bite and then gastroscopy was performed.The ordinary endoscopic bite group began to perform endoscopic operation after sufficient sedation was achieved.In both groups, 5mg/kg·h propofol was injected continuously to maintain anesthesia until the examination was completed.If participants showed frowning or slight body movement during diagnosis and treatment, 40 to 50mg of propofol was added intravenously.If HR < 50 times/intravenous injection of atropine 0.5mg;MAP < 60mmHg intravenous hydroxyamine 1mg;When SpO2 < 92%, artificial airway intervention such as jaw support, assisted breathing or mask was given.After the examination, study participants were not allowed to leave the examination room until they had a MOAA/S score of 3-4.If the sedation/anaesthesia Discharge rating scale scores more than 9 points, patients can be accompanied by relatives and friends.The incidence of hypoxia (75%≤SpO2 < 90%, ≤60s) and severe hypoxia (SpO2 < 75% or 75%≤SpO2 < 90%, ≥60s) during anesthesia were recorded.The incidence of choking, reflux aspiration and laryngeal spasm were recorded.The time of intervention was half or disappearance of end-expiratory carbon dioxide and/or disappearance of thoracic fluctuation and/or SpO2 < 95%, that is, opening the airway successively until SpO2≥95%, and recording the last means of opening the airway.The means of opening the airway of the two groups were the same, including: 1) adjusting the oxygen flow;2) Lift the lower jaw;3) Mask ventilation (pull out the gastroscope if necessary);4) Tracheal intubation or laryngeal mask for ventilator assisted ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* 30≤BMI≤40
* Written informed consent of patient or family
* painless stomach + colonoscopy
* ASA grade I-II

Exclusion Criteria：

* Patients with blood clotting disorders or a tendency to oropharyngeal bleeding, mucosal damage or space occupation, difficulty in placing oropharyngeal airway, etc., who cannot perform oropharyngeal airway ventilation;
* Severe cardiac insufficiency (≤4mets);
* Patients with severe renal insufficiency;
* diagnosed severe hepatic insufficiency;
* Diagnosed with chronic obstructive pulmonary disease (COPD) or currently suffering from other acute or chronic lung diseases, requiring long-term or intermittent oxygen therapy;
* Increased intracranial pressure;
* Upper respiratory tract infections such as mouth, nose or throat;
* Fever (core body temperature ≥37.5℃);
* A confirmed diagnosis of pregnancy or breastfeeding;
* Allergic to sedatives such as propofol or equipment such as tape;
* Emergency surgery;
* Multiple trauma;
* SpO2 < 95% before operation;
* A history of drug and/or alcohol abuse within 2 years prior to the start of the screening period;(Drinking more than three times standard alcoholic beverages per day, equivalent to about 10g of alcohol or equivalent to 50g of Chinese liquor);
* Patients with previous psychiatric and neurological diseases, such as depression, severe central nervous depression, Parkinson's disease, basal ganglia disease, schizophrenia, epilepsy, Alzheimer's disease, myasthenia gravis;
* Currently participating in other clinical trials;
* Patients who are deemed unfit by the investigator to participate in the trial;
* Patients with a history of smoking were excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxia | 1 minute after anesthesia induction
  To investigate the incidence of new oropharyngeal airway hypoxia (75%≤SpO2 < 90%, ≤60s) during anesthesia in patients undergoing painless gastroenteroscopy

SECONDARY OUTCOMES:
The incidence of severe hypoxia | 1 minute after anesthesia induction
  The incidence of severe hypoxia (SpO2 < 75% or 75% ≤SpO2 < 90%, ≥60s)
The incidence of requiring airway intervention | 1 minute after anesthesia induction
  Serious adverse events such as tracheal intubation, non-invasive ventilation are required
The dosage of additional drugs was recorded during the operation | 1 minute after anesthesia induction
  The dosage of additional drugs was recorded during the operation
The satisfaction of endoscopists was recorded | Within 30 minutes after anesthesia awakening
  The doctor satisfaction rating scale also uses a 0-10 rating scale, where 0 represents very dissatisfied and 10 represents very satisfied. Endoscopes need to select a corresponding number on the scoring table based on their actual experience to indicate whether the patient is satisfied with the patient's cooperation and response to the operation process.
Recorded adverse events | 1 minute after anesthesia induction
  The incidence of choking, laryngeal spasm and reflux aspiration were observed.Apnea or slow breathing episodes (defined as respiratory rate ≤6 beats/min);Bradycardia is defined as a heart rate ≤50 beats/min.Serious adverse events such as tracheal intubation, non-invasive ventilation, use of vasopressors, and hospitalization are required.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Wu, Principal Investigator — Department director

IPD SHARING:
Plan to Share IPD: No